CLINICAL TRIAL: NCT04717024
Title: The Nanowear Wearable Covid-19 Observational and Analysis Trend
Acronym: NanoCOAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanowear Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NWCT20-SS-002
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Observational Study - no intervention — Observational Study - no intervention

SUMMARY:
The NanoCOAT study is a multi-center, prospective, non-randomized, feasibility, observational, non-significant risk study. The NanoCOAT study will enroll a minimum of 10 and a maximum of 100 subjects in a potential for a multi-site in order to collect data and analyze physiological and biometric trends due to Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Male or female over the age of 18 years
* The patient is currently hospitalized with a primary diagnosis of Covid-19

Exclusion Criteria:

* Subject is unwilling or unable to wear the vest during hospitalization.
* Subjects who are pregnant.
* Subject is intubated or admitted to ICU
* Subject has an implantable cardiac device (i.e pacemaker or internal cardioverter defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of legal age to give informed consent who are currently or recently hospitalized with a primary diagnosis of Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hosptialized patient data | up to 30 days of monitoring leading to discharge or admission to ICU
  The primary study endpoint is adequate collection of hospitalized COVID 19 patient health metric data through the Nanowear WMDRS

SECONDARY OUTCOMES:
Trends in COVID 19 exacerbation | up to 30 days of monitoring leading to discharge or admission to ICU
  Exploratory information will be used to compare the signals obtained from the device to the severity of Covid-19 as measured by clinical evaluation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Maimonides Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No